CLINICAL TRIAL: NCT03781245
Title: Integrated Approaches to Health and Safety in a Dynamic Construction Work Environment (All the Right Moves for Subcontractors)
Brief Title: Integrated Approaches to Health and Safety in a Dynamic Construction Work Environment
Acronym: ARM For SUBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Jack Dennerlein, Associate Director, Center for Work, Health, & Well-being, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB13-1948
Record Dates: First submitted 2018-11-20; First posted 2018-12-19 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Worker Health; Work Injury; Safety Climate; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early (Experimental): Intervention is administered for cycle 1 and 2 with researchers and following this the company continues intervention independently.
  Interventions: Other: All the Right Moves for Subcontractors
- Lagged (Active Comparator): Intervention is not administered for cycle 1; researchers administer intervention in cycle 2 and following this the company continues intervention independently.
  Interventions: Other: All the Right Moves for Subcontractors

INTERVENTIONS:
Other: All the Right Moves for Subcontractors — "All the Right Moves for Subcontractors" aims to improve safety, health and wellbeing, through the development of a communication infrastructure with supplemental tools where construction workers and company mangers work together to collaboratively identify problems and strategies to improve their conditions of work. The intervention is grounded in the key characteristics of integrated organizational interventions to improve workers' health safety and wellbeing detailed in Harvard Center for Work, Health and Wellbeing's Implementation Guidelines (McLellan et al, 2016).
  The intervention involves a cyclical approach through which the research team facilitate a participatory process to identify workers' health concerns, prioritize these concerns, use an action planning process to identify and operationalize solutions, and develop a company-specific evaluation plan to measure change.
  Other Names: ARM for SUBS

SUMMARY:
"All the Right Moves for Subcontractors" aims to improve safety, health and well-being, through the development of a communication infrastructure with supplemental tools where construction workers and company mangers (project, operations and safety) work together to collaboratively identify problems and strategies to improve their conditions of work. The intervention is grounded in the key characteristics of integrated organizational interventions to improve workers' health safety and well-being detailed in Harvard Center for Work, Health and Well-being's Implementation Guidelines (McLellan et al, 2016).

The intervention involves a cyclical approach through which the research team facilitate a participatory process to identify workers' health concerns, prioritize these concerns, use an action planning process to identify and operationalize solutions, and develop a company-specific evaluation plan to measure change. We will evaluate this program by measuring safety climate, health climate, pain and injury and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* All workers employed by the recruited contractors at the eligible worksites

Exclusion Criteria:

* Companies with less than 5 workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Worker Outcomes: Injury assessed by the Nordic Musculoskeletal Questionnaire | Change from Baseline at 2 months, 4 months, and 6 months
  NMQ has been applied to a wide range of occupational groups to evaluate musculoskeletal problems Scale:0-1 0:minimum
  1:maximum
Worker Outcomes: Pain assessed by the Nordic Musculoskeletal Questionnaire | Change from Baseline at 2 months, 4 months, and 6 months
  NMQ has been applied to a wide range of occupational groups to evaluate musculoskeletal problems Scale:0-1 0:minimum
  1:maximum
Enterprise Outcomes: Work Productivity and Activity Impairment assessed by Work Productivity and Activity Impairment Questionnaire (WPAI) | Change from Baseline at 2 months, 4 months, and 6 months
  Work Productivity and Activity Impairment Questionnaire (WPAI) measures impairment due to the specified problem and all health problems.
  Scale:0-1 0:minimum
  1:maximum
Enterprise Outcomes: Health Climate assessed by questions modified from safety climate scale for construction workers | Change from Baseline at 2 months, 4 months, and 6 months
  Questions adapted from safety climate scale: Jorgensen, E., Sokas, R. K., Nickels, L., Gao, W., & Gittleman, J. L. (2007). An English/Spanish safety climate scale for construction workers. American journal of industrial medicine, 50(6), 438-442.
  Scale:0-1 0:minimum
  1:maximum
Enterprise Outcomes: Safety Climate assessed by using the validated scale: An English/Spanish safety climate scale for construction workers. | Change from Baseline at 2 months, 4 months, and 6 months
  Jorgensen, E., Sokas, R. K., Nickels, L., Gao, W., & Gittleman, J. L. (2007). An English/Spanish safety climate scale for construction workers. American journal of industrial medicine, 50(6), 438-442.
  Scale:0-1 0:minimum
  1:maximum

SECONDARY OUTCOMES:
Worker Health Behaviors: Diet | Change from Baseline at 2 months, 4 months, and 6 months
  PrimeScreen Questionnaire; Rifas-Shiman SL, Willett WC, Lobb R, Kotch J, Dart C, Gillman MW. PrimeScreen, a brief dietary screening tool: reproducibility and comparability with both a longer food frequency questionnaire and biomarkers. Public Health Nutr. 2001 Apr;4(2):249-54 Scale: 0-4 0:minimum 4:maximum
Worker Health Behaviors: Leisure Physical Activity | Change from Baseline at 2 months, 4 months, and 6 months
  International Physical Activity Questionnaire (Short Form)http://uacc.arizona.edu/sites/default/files/ipaq_english_telephone_short.pdf Scale: 0-7 days 0=minimum 7=maximum
Worker Health Behaviors: Alcohol Use assessed by using validated questions from NIAAA | Change from Baseline at 2 months, 4 months, and 6 months
  National Institute on Alcohol Abuse and Alcoholism Scale:0-9 0:minimum 9:maximum https://www.niaaa.nih.gov/research/guidelines-and-resources/recommended-alcohol-questions
Worker Health Behaviors: Tobacco Use assessed by modifying questions from the National Adult Tobacco Survey (NATS) | Change from Baseline at 2 months, 4 months, and 6 months
  Dichotomous questions adapted from the National Adult Tobacco Survey (NATS) Scale:0-2 0:minimum 2:maximum
Psychosocial Work Environment: Co-worker Support assessed by assessed by Job Content Questionnaire (JCQ), a validated scale. | Change from Baseline at 2 months, 4 months, and 6 months
  Uses questions from the Job Content Questionnaire (JCQ), a validated scale by Karasek_et_al__1998 Scale:0-1 0:minimum
  1:maximum
Psychosocial Work Environment: Supervisor Support assessed by Job Content Questionnaire (JCQ), a validated scale. | Change from Baseline at 2 months, 4 months, and 6 months
  Uses questions from the Job Content Questionnaire (JCQ), a validated scale by Karasek_et_al__1998 Scale:0-1 0:minimum
  1:maximum
Psychosocial Work Environment: Communication assessed by Job Content Questionnaire (JCQ), a validated scale. | Change from Baseline at 2 months, 4 months, and 6 months
  Uses questions from the Job Content Questionnaire (JCQ), a validated scale by Karasek_et_al__1998 Scale:0-1 0:minimum
  1:maximum

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters SE, Trieu HD, Manjourides J, Katz JN, Dennerlein JT. Designing a Participatory Total Worker Health(R) Organizational Intervention for Commercial Construction Subcontractors to Improve Worker Safety, Health, and Well-Being: The "ARM for Subs" Trial. Int J Environ Res Public Health. 2020 Jul 15;17(14):5093. doi: 10.3390/ijerph17145093. PMID 32679687
- See also: Implementing an Integrated Approach Weaving Worker Health, Safety, and Well-being into the Fabric of Your Organization. — http://centerforworkhealth.sph.harvard.edu/sites/default/files/10.12.17_Guidelines_Screen_post.pdf